CLINICAL TRIAL: NCT04986501
Title: Clinical Evaluation of MucoPEG™ for Xerostomia
Acronym: CEMPEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SunBio, Inc. (Industry)
Collaborators: NAMSA (Other); Rudacure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SB-MU-001
Record Dates: First submitted 2021-07-08; First posted 2021-08-02 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-06

CONDITIONS: Dry Mouth; Xerostomia
Keywords: Dry mouth; Xerostomia; Cotton mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: The study is a randomized, open-labelled crossover trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MucoPEG (Experimental): Arm being compared to against Biotene
  Interventions: Device: MucoPEG
- Biotene (Active Comparator): Arm being compared against MucoPEG
  Interventions: Device: Biotene

INTERVENTIONS:
Device: MucoPEG — Experimental
  Arms: MucoPEG
Device: Biotene — Active Comparator
  Arms: Biotene

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the oral rinse comparing to MucoPEG™ and Biotene®.

This is a randomized open-label crossover study with 42 patients receiving treatment. Patients will be randomly assigned to receive either the MucoPEG™ or the Biotene® Dry Mouth Gentle Oral Rinse in the first period. Patients will use the assigned oral rinse two times a day for two weeks. Patients will switch to the other treatment after a wash-out period of one week.

DETAILED DESCRIPTION:
The purpose of this study is to compare MucoPEG™ and it temporal change to those of the Biotene® Dry Mouth Gentle Oral Rinse in patients with Xerostomia. The study will gather data on patient reported outcomes on the safety and performance of the product, mouth-feel qualities and any changes in dry mouth.

ELIGIBILITY:
Inclusion Criteria:

1. Must have read, understood and signed an informed consent prior to entering the study.
2. Must be 18 years of age or older
3. Good general and mental health with, in the opinion of the investigator or their medically qualified designee, no clinically relevant or significant abnormalities found on examination of the oral cavity or in their medical history.
4. Participant with a Challacombe Scale score of 1 or higher
5. Participant agrees not to eat, drink, chew tobacco, chew gum, smoke, brush or floss their teeth for 2 hours prior to study visits
6. Participant agrees not to use any oral care products or any type of breath mint or lozenges for 2 hours prior to study visits
7. Participant agrees not to consume any food or liquid during the study visits, except for what is provided by the study research staff (e.g., water and treatments A and B during evaluation periods)
8. Participant agrees to using clinical oral care supplies provided by the investigators and no other products during the entire study
9. Understands and is willing and able to comply with all study procedures and restrictions

Exclusion Criteria:

1. Women who are pregnant or intending to become pregnant over the course of the study, or who are found to have a positive urine pregnancy test at the Screening Visit
2. Women who are breast-feeding
3. Participant is currently undergoing radiotherapy and/or chemotherapy.
4. Any condition the investigator identifies that may impede the participant's ability to properly participate in the study. For example, Alzheimer's Disease
5. Participant with untreated oral mucosal disease which in the opinion of the investigator could interfere with the study. For example, presence of oral ulceration.
6. Evidence of gross intra-oral neglect or need for extensive dental therapy
7. Denture wearer (complete dentures)
8. Participant on systemic parasympathetic medications (e.g. pilocarpine) for treating dry mouth, but the dose requirement of which is unstable
9. Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or to any of their stated ingredients
10. Participation in another clinical study (including studies of cosmetic products) or in receipt of an investigational drug within 14 days of the screening visit
11. Previous participation in this study
12. Recent history (within one year prior to screening visit) of alcohol or other substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: To be determined To be determined, DDS, Principal Investigator — Study Site
Locations (2):
- United States (2):
  - ColoradoENT, Colorado Springs, Colorado
  - Tufts University School of Dental Medicine, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study prospectively enrolled 45 subjects from 2 investigational sites across the USA starting 3 MAY 2022.
  Twenty-two subjects were enrolled, with twenty-one completing the study at Tufts University School of Dental Medicine in Boston, MA, over approximately 42 days.
  Twenty-three subjects were enrolled, with twenty-one completing the study at Colorado ENT & Allergy in Colorado Springs, CO.
Pre-assignment Details: 42 subjects were randomized. 3 subjects were not randomized. why the subjects (n = 3) exited the study early, were screen failure, withdrawal of consent, and lost of follow-up before randomization.
Groups:
- MucoPEG First, Then Biotène®: Participants first used MucoPEG two times a day, once after breakfast and once before bedtime for 2 weeks. After a washout period of 1 weeks, they then used Biotene two times a day for 2 weeks.
- BIotene First, Then MucoPEG: Participants first used Biotene two times a day for 2 weeks. After a washout period of 1 weeks, they then used MucoPEG two times a day, once after breakfast and once before bedtime for 2 weeks.
Period: First Intervention(2 Weeks)
Arm/Group | MucoPEG First, Then Biotène® | BIotene First, Then MucoPEG
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0
Period: Second Intervention(2 Weeks)
Arm/Group | MucoPEG First, Then Biotène® | BIotene First, Then MucoPEG
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients will be randomly allocated to either group A or group B in this crossover study in a 1:1 ratio. Patients in group A will begin using MucoPEG from Visit 2 for two weeks (period 1). This is followed by a washout period of one week. They will switch to using Biotène® Dry Mouth Gentle Oral Rinse from Visit 5 for another two weeks (period 2). Patients in group B will follow the same pattern except they receive Biotène® Dry Mouth Gentle Oral Rinse in period 1 and MucoPEG in period 2.
Groups:
- All Study Participants: Participant will be randomly allocated to either MucoPEG or Biotene in this crossover study in a 1:1 ratio. Participants first received MucoPEG or Biotene for 2 weeks. After a washout period of 1 weeks, they then received Biotene or MucoPEG for 2 weeks.
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42
Challacombe Scale Score [Mean (Standard Deviation); unit: units on a scale] — The Challacombe Scale works as an additive score of 1 to 10.
  1 being the least and 10 being the most severe. Each feature scores 1 and symptoms will not necessarily progress in the order shown, but summated scores indicate likely patient needs. Score changes over time can be used to monitor symptom progression or regression.
  units on a scale | 3.3 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in VAS for Mouth Dryness
Description: To demonstrate the effectiveness of MucoPEG is better than that of Biotene Dry Mouth Gentle Oral Rinse in relieving xerostomia. Effectiveness will be addressed using the Visual Analogue Scale (VAS). (VAS), where 0 is "Not Dry at All" and 10 is "Very Dry" VAS (before), which is measured before using any of the products on the first day of each treatment period, at Visit 2 or Visit 5. VAS (end), which is measured after the last dose of a product on the final day of each treatment period, at Visit 4 or Visit 7.
  Change in the rating of mouth dryness is the difference between the two time points, that is, VAS (end) - VAS (before).
Time Frame: baseline and 2 weeks, value at 2weeks minus value at baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MucoPEG | Biotene
Number analyzed (Participants) | 42 | 42
score on a scale
  Period 1: number analyzed (Participants) | 20 | 22
  Period 1 | -0.8 (2.0) | -0.7 (3.0)
  Period 2: number analyzed (Participants) | 22 | 20
  Period 2 | -1.5 (2.4) | -0.4 (1.6)
Statistical Analysis 1: Comparison: MucoPEG vs Biotene; Test type: Superiority; p < 0.01, t-test, 1 sided

2. Primary Outcome: Dry Mouth Relief Questionnaires (DMRQ)
Description: The effect of MucoPEG™ in relieving xerostomia, relative to that of Biotène was assessed using the Dry Mouth Relief Questionnaires (DMRQ). This questionnaire was given to the patients to answer the following question: "Does the product relieve the discomfort of dry mouth?" To answer the question, only one of the answer options is selected: 1. None/ (No Relief), 2. Not Enough, 3. Some/ Good, 4. Very Good, 5. Significant/ Excellent A favorable responses on the Dry Mouth Relief Questionnaire (DMRQ) include "4 - very good" or "5 - significant/excellent." The numbers are the number of patients who responded favorably at their last visit.
Time Frame: 2 weeks(at last visit)
Population: as for baseline characteristics
Measure: Number; unit: participants response with 4 or 5 score
Arm/Group | MucoPEG | Biotene
Number analyzed (Participants) | 42 | 42
participants response with 4 or 5 score | 10 | 11

3. Primary Outcome: Change in VAS for Tongue Dryness
Description: as for outcome 1
Time Frame: baseline and 2 weeks, value at 2weeks minus value at baseline
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MucoPEG | Biotene
Number analyzed (Participants) | 42 | 42
score on a scale
  Period 1: number analyzed (Participants) | 20 | 22
  Period 1 | -0.6 (2.4) | -0.4 (3.3)
  Period 2: number analyzed (Participants) | 22 | 20
  Period 2 | -1.4 (2.4) | -0.2 (1.3)
Statistical Analysis 1: Comparison: MucoPEG vs Biotene; Test type: Superiority; p < 0.01, t-test, 1 sided

4. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Evaluated by the Principal Investigator
Description: To evaluate the clinical safety of MucoPEG. Patient reported outcomes will be evaluated by the Principal Investigator.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MucoPEG | Biotene
Number analyzed (Participants) | 42 | 42
Participants | 0 | 0

5. Secondary Outcome: Dry Mouth Inventory (DMI) Questionnaire.
Description: To demonstrate the effectiveness using the Dry Mouth Inventory (DMI). There are 8 Dry Mouth Inventory (DMI) questionaires as follows. 1. My mouth feels dry, 2. I have difficulty eating dry foods, 3. I get up at night to drink, 4. My mouth feels dry when eating a meal, 5. I sip liquids to aid in swallowing food, 6. I suck sweets or cough lollies to relieve dry mouth, 7. My lips stick to the teeth, 8. My tongue sticks to the roof of my mouth.
  Using a scale from "Disagree (0)" to "Strongly agree (3)". The scale has a minimum value of "0" and a maximum value of "24". The larger the scale, the more severe the dry mouth.
Time Frame: 2 weeks
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MucoPEG | Biotene
Number analyzed (Participants) | 42 | 42
score on a scale | 9.4 (5.3) | 9.4 (5.6)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at treatment period (35days)
Arm/Group | MucoPEG | Biotene
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 1/42 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MucoPEG (N=42) | Biotene (N=42)
celiac disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food reaction (General disorders) | 1 (1) | 0 (0)
sinus infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT04986501/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT04986501/SAP_001.pdf